CLINICAL TRIAL: NCT01799772
Title: The Feasibility of a Comprehensive Behavioral Intervention in Patient Post Total Knee Arthroplasty
Brief Title: The Feasibility of a Comprehensive Behavioral Intervention in Patient Post TKA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO11030404
Record Dates: First submitted 2013-02-08; First posted 2013-02-27 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Comprehensive behavioral intervention (Experimental): It will involve regular contacts over 6 month period. It will include 2 weekly contacts for weeks 1-6, weekly contacts for weeks 7-8, bi-weekly contact for months 3-4, and monthly contact for months 5-6. There is a combination of 20 individual and group-based sessions.
  It is a combination of 4 components: a) Evidence-based exercise program, b) Physical activity promotion, c) Healthy nutrition guidance, and d) Self-management.
  Interventions: Behavioral: Comprehensive Behavioral Intervention
- Standard of Care Exercise Program (SCE) (Active Comparator): The SCE will be delivered by a physical therapist. It represents the typical rehabilitation after TKA surgery. It is expected to provide small and short-lived functional improvement. Subjects will participate in 12 supervised sessions (2 x/week, for 6 weeks). The SCE consists of: a) lower extremity range of motion and stretching exercises, b) lower extremity strengthening exercises of moderate intensity, and d) endurance exercises using treadmill.
  Interventions: Other: Standard of Care Exercise Program

INTERVENTIONS:
Behavioral: Comprehensive Behavioral Intervention — 1. Evidence-based exercise program - Combination of high intensity lower extremity strengthening, endurance on the treadmill, functional task-oriented exercises, and balance techniques. During 12 sessions, subjects will be instructed to become independent in performing the exercises at home.
  2. Physical activity promotion - Instructions to engage in moderate intensity exercise 5 days/week will be delivered along with the exercise program.
  3. Healthy nutrition guidance - Instructions on healthy nutrition delivered by a dietitian.
  4. Self-management - Basic self-management skills advocated by the Arthritis Foundation Self-Help Program and behavioral strategies (self-monitoring, problem solving, relapse prevention, and goal-setting) and feedback into approaches a, b and c.
  Arms: Comprehensive behavioral intervention
Other: Standard of Care Exercise Program — Typical rehabilitation after TKA surgery
  Arms: Standard of Care Exercise Program (SCE)

SUMMARY:
Patients who undergo a replacement of their knees are generally older adults who have dealt with severe knee pain and joint degeneration for a long time. The majority of them are sedentary, and around 1/3 are obese. The knee replacement surgery decreases knee pain and helps patients to live a better life. However, after the surgery, some patients have difficulty performing basic activities such as walking, or going up-down stairs, and the majority remains sedentary and gain weight. These combined problems leave patients at risk of worsening their health. Therefore, a treatment that takes care of all these combined problems is needed. We propose an all-inclusive treatment, called comprehensive behavioral intervention (CBI) that intends to improve the long-term effects of exercise programs. The CBI combines exercise program with promotion of physical activity, orientation on healthy nutrition, and an education approach that promotes self-initiative towards healthy habits. The overall aim of this proposed study is to test how patients post TKA will like the CBI program, how safe the program is, and adapt the program as needed for better acceptability. We believe the CBI will be safe, well tolerated, and will improve the ability of patients to perform physical tasks. We also believe the program will increase the amount of physical activity, will promote maintenance of healthy weight, and will help the patients to obtain and maintain healthy habits. In this study subjects will be selected by a flip of a coin to receive either our CBI program or a more traditional exercise program. Subjects will be tested before and after the treatments. Our measures of main interest are how well subjects move around and how physically active they are. We are also interested on the effect of the interventions on body weight, blood pressure, eating habits, and general health. The team of researchers for this study includes several disciplines. The proposed study will defend the need for a larger study that can have a very important impact on the public health of patients post TKA. The reason for the public health impact is if the physical limitations experiences by patients post TKA are left untreated, they tend to get worse. Furthermore, by increasing physical activity and promoting healthy weight, it may improve general health and prevent chronic diseases. Last, developing educational intervention that promotes self-initiative will result in long-term health benefits post TKA.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral TKA at least three months prior to, but no longer than six months prior to study participation;
* Surgical technique was a minimally invasive (quadriceps sparing) TKA performed by the same experienced surgeon;
* Provide a written medical clearance to participate in the study;
* Speak fluent English;
* Are older than 50 years.

Exclusion Criteria:

* Have bilateral or TKA revision;
* Have hip or ankle joint replacement;
* Are unable to comfortably bear weight on the surgical knee;
* Had 2 or more falls within past year;
* Have uncontrolled medical condition that would prevent safe participation in the study (uncontrolled blood pressure, dyspnea at rest, cardiovascular disease, absolute contraindications to exercise, and diabetes);
* Participating in regular exercise during prior 6 months;
* Use beta blockers,
* Have a neurological condition that affects locomotion;
* Have had a malignancy, life-threatening illness or surgery in the past six months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Self-reported physical function | 6 months
  Change from Baseline in Western Ontario and McMaster Universities Osteoarthritis Index - Physical Function scale (WOMAC-PF) at 6 months.

SECONDARY OUTCOMES:
Change from Baseline in Performance-based physical function | 6 months
  Change from Baseline in Self-selected gait speed at 6 months.
Change from Baseline in Performance-based Physical Function | 6 months
  Change from Baseline in Timed 5 chair rise at 6 months.
Change from Baseline in Performance-based Physical Function | 6 months
  Change from Baseline in single leg balance time at 6 months.
Change from Baseline in Performance-based Physical Function | 6 months
  Change from Baseline in timed ascend/descend stair test at 6 months.
Change from Baseline in Performance-based Physical Test | 6 months
  Change from Baseline in 6 minutes walk test at 6 months.

OTHER OUTCOMES:
Change from Baseline in measures of physical activity | 6 months
  Change from Baseline in measures of physical activity taken by a portable activity monitor at 6 months.
Change from Baseline in measures of General Health Status | 6 months
  Change from Baseline in the Medical Outcomes Survey 36-Item Short-Form Health Survey at 6 months.
Change from Baseline in measures of physical activity | 6 months
  Change from Baseline in measures of physical activity taken by a self-reported questionnaire (CHAMPS) at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Sara R Piva, PT, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Piva SR, Almeida GJ, Gil AB, DiGioia AM, Helsel DL, Sowa GA. Effect of Comprehensive Behavioral and Exercise Intervention on Physical Function and Activity Participation After Total Knee Replacement: A Pilot Randomized Study. Arthritis Care Res (Hoboken). 2017 Dec;69(12):1855-1862. doi: 10.1002/acr.23227. Epub 2017 Nov 2. PMID 28217891